CLINICAL TRIAL: NCT05180240
Title: Impact of CardiolRx on Myocardial Recovery in Acute Myocarditis. A Double-blind, Placebo-controlled Trial
Brief Title: Impact of CardiolRx on Myocardial Recovery in Patients With Acute Myocarditis
Acronym: ARCHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiol Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cardiol 100-002
Record Dates: First submitted 2021-09-25; First posted 2022-01-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Myocarditis
Keywords: Pharmaceutically produced CBC; THC < 5ppm
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Multi-center, double-blind, randomized, placebo-controlled, parallel group design. 1:1 randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo will match active study drug in color, odor, taste and appearance to assure proper blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CardiolRx (Experimental): * Week 1 (p.m. dose of Day 1 to a.m. dose of Day 7): 2.5 mg/kg of body weight b.i.d. CardiolRxTM or placebo
  * Week 2 (p.m. dose of Day 7 to a.m. dose of Day 14): 5 mg/kg of body weight b.i.d. CardiolRxTM or placebo
  * Week 3 (p.m. dose of Day 14 to a.m. dose of Day 21): 7.5 mg/kg of body weight b.i.d. CardiolRxTM or placebo
  * Week 4 to end of treatment period (p.m. dose of Day 21 to a.m. dose of last day of treatment period at week 12): 10 mg/kg of body weight b.i.d. CardiolRxTM or placebo
  Interventions: Drug: CardiolRx
- Placebo (Placebo Comparator): * Week 1 (p.m. dose of Day 1 to a.m. dose of Day 7): 2.5 mg/kg of body weight b.i.d. CardiolRxTM or placebo
  * Week 2 (p.m. dose of Day 7 to a.m. dose of Day 14): 5 mg/kg of body weight b.i.d. CardiolRxTM or placebo
  * Week 3 (p.m. dose of Day 14 to a.m. dose of Day 21): 7.5 mg/kg of body weight b.i.d. CardiolRxTM or placebo
  * Week 4 to end of treatment period (p.m. dose of Day 21 to a.m. dose of last day of treatment period at week 12): 10 mg/kg of body weight b.i.d. CardiolRxTM or placebo
  Interventions: Drug: CardiolRx

INTERVENTIONS:
Drug: CardiolRx — Eligible patients will be randomized to receive CardiolRx or placebo. Intervention will be administered orally (via syringe) with food twice daily.
  Other Names: Cannabidiol

SUMMARY:
Multi-center, double-blind, placebo-controlled, parallel group design. Patients with myocarditis will be screened and, if eligible, randomized within 10 days of the diagnostic CMR to CardiolRx or placebo.

CardiolRx is pharmaceutically produced Cannabidiol and is free of tetrahydrocannabinol (THC<5 ppm). The treatment period is 12 weeks; a last follow-up visit is scheduled one week after the last treatment, 13 weeks after randomization. Study assessments include Cardiac Magnetic Resonance imaging (CMR), ECG monitoring, the Kansas City Cardiomyopathy Questionnaire (KCCQ), the Columbia-Suicide Severity Rating Scale (C-SSRS) as well as physical exams and laboratory tests.

The primary and secondary outcome parameters are measured by CMR. Additional outcomes include clinical endpoints and changes in inflammatory and biomarkers.

DETAILED DESCRIPTION:
Rationale:

Myocarditis is an acute inflammatory condition of the myocardium. Presentation of the disease may be fulminant and necessitate cardiac support, or even result in sudden cardiac death; milder cases are usually self-limiting but may progress to dilated cardiomyopathy with eventual end-stage heart failure. Other than treatments for associated heart failure there are no specific indicated treatments for myocarditis. CardiolRxTM (cannabidiol [CBD] solution), which is known to have anti-inflammatory properties, is being investigated to treat the underlying inflammatory process and thereby favorably modify acute myocarditis. The primary endpoints of the trial are cardiac magnetic resonance measures of left ventricular systolic function (ejection fraction and longitudinal strain) and myocardial edema (extra cellular volume) which have been shown to predict long term prognosis of patients with acute myocarditis.

Multi-center, double-blind, randomized, placebo-controlled, parallel group design. 1:1 randomization; treatment will be stratified within sites.

Patients diagnosed with acute myocarditis by a biopsy or a CMR will be screened within 10 days of the diagnostic CMR. Informed consent will be obtained at this point. For patients who have been diagnosed using an EMB, a CMR needs to be performed as well, which will be included in the informed consent form (ICF).Eligible patients will then be randomized within 10 days from the CMR assessment.

Baseline assessments include the following: Clinical assessment, including vital signs, ECG, 24-hr Holter, chest x-ray; Hematology and blood chemistry, NYHA classification, C SSRS and KCCQ. Frozen plasma will be retained for central analysis of hs-troponin, NT-proBNP and inflammatory markers.

Study treatment needs to be taken with food and will be initiated in the evening of Day 1, after all baseline assessments have been completed and the patient has been randomized.

Oral administration is as follows:

• Week 1 (p.m. dose of Day 1 to a.m. dose of Day 7): 2.5 mg/kg of body weight b.i.d. CardiolRxTM or placebo

* Week 2 (p.m. dose of Day 7 to a.m. dose of Day 14):

  5 mg/kg of body weight b.i.d. CardiolRxTM or placebo
* Week 3 (p.m. dose of Day 14 to a.m. dose of Day 21):

7.5 mg/kg of body weight b.i.d. CardiolRxTM or placebo • Week 4 to end of treatment period (p.m. dose of Day 21 to

a.m. dose of last day of treatment period at week 12): 10 mg/kg of body weight b.i.d. CardiolRxTM or placebo

If the next higher dose after each study drug increase is not tolerated, the dose will be reduced to the previous tolerated dose.

Every week (before the next dose increase) the patient will be re-evaluated. This includes ECG monitoring at approximately 5 hours post-morning dose (time of Tmax) to surveil for deleterious effects on ECG intervals (particularly the QTc interval) and rhythm. Drug titration will be dependent on investigator or designate interrogation of the ECGs and the absence of new, clinically significant abnormalities on those ECGs.

Vital signs, concurrent medication and Adverse Events (AEs), including Serious Adverse Events (SAEs) will be recorded, blood chemistry including liver function tests, hematology as well as INR assessments will be carried out.

Final efficacy assessments (including a second CMR) will take place after 12 weeks of study treatment. A final safety assessment will take place after 13 weeks, 1 week after completion of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older
2. Diagnosed with acute myocarditis including:

   1. Clinical criteria (symptoms of chest pain, arrhythmia or shortness of breath, or history of viral-like illness), preferably followed by elevated troponin PLUS
   2. CMR diagnosis (Lake Louise Criteria) within 10 days prior to randomization OR
   3. Endomyocardial biopsy (EMB) showing either cellular inflammation and/or immunohistochemistry consistent with inflammation.
3. Male subjects with partners of childbearing potential who have had a vasectomy or are willing to use double barrier contraception methods during the conduct of the study and for 2 months after the last dose of study drug.
4. Women of childbearing potential willing to use an acceptable method of contraception starting with study drug administration and for a minimum of 2 months after study completion. Otherwise, women must be post- menopausal.

Exclusion Criteria:

1. Coronary artery disease (CAD) defined as a stenosis greater than 50% in a major epicardial coronary artery
2. Severe valvular heart disease
3. Inability to safely undergo CMR including administration of gadolinium
4. Estimated glomerular filtration rate (eGFR) < 30 ml/min
5. Elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal (ULN) or ALT or AST >3x ULN plus bilirubin >2x ULN.
6. Sepsis, defined as documented bacteremia at the time of presentation or other documented active infection.
7. Severe left ventricular (LV) dysfunction requiring inotropic support, left ventricular assist device (LVAD) or other circulatory assist devices, or urgent need for transplantation
8. Documented biopsy evidence of giant cell or eosinophilic myocarditis
9. Prior history of sustained ventricular arrhythmia
10. Acute coronary syndrome within 30 days
11. Percutaneous coronary intervention within 30 days
12. History of QT interval prolongation or QTc interval > 500 msec
13. Treated with strong inducers CYP3A4 or CYP2C19, as listed in Appendix 17.8
14. Treated with digoxin and/or type 1 or 3 antiarrhythmics
15. Current participation in any research study involving investigational drugs or devices
16. Inability or unwillingness to give informed consent
17. Ongoing drug or alcohol abuse
18. Women who are pregnant or breastfeeding
19. Current diagnosis of cancer, with the exception of non-melanoma skin cancer
20. Any factor, which would make it unlikely that the patient can comply with the study procedures
21. On any cannabinoid during the past month
22. Body weight > 170 kg
23. Showing suicidal tendency as per the C-SSRS, administered at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
extracellular volume (ECV) | 12 weeks post randomization
  primary
Global longitudinal Strain (GLS) | 12 weeks post randomization
  primary

SECONDARY OUTCOMES:
Left-ventricular ejection fraction (LVEF) | 12 weeks post randomization
  secondary endpoint

OTHER OUTCOMES:
Percentage of patients recovered | From baseline to 12 weeks of treatment
  defined as LVEF ≥ 0.55 at 12 weeks of treatment
Survival, free from major event | 12 weeks post randomization
  Major event defined as cardiac transplant, left-ventricular assist device (LVAD), hospitalization for Heart failure (HF)
Change in CMR parameters (%) | From baseline to 12 weeks of treatment
  Any change in CMR parameters from baseline to 12 weeks post randomization:
  LVEF (%), ECV (%), GLS (%), LGE (%)
Change in CMR parameters (mL/m2) | From baseline to 12 weeks of treatment
  Any change in CMR parameters from baseline to 12 weeks post randomization:
  LVEDV (ml/m2), LVESV (ml/m2), LAESV (ml/m2).
Change in CMR parameters (g/m2) | From baseline to 12 weeks of treatment
  Any change in CMR parameters from baseline to 12 weeks post randomization:
  LV mass (g/m2)
New York Heart Association classification (NYHA) | From baseline to 12 weeks of treatment
  New York Heart Association classification (NYHA) ranked in order of best to worse outcome from Class I (best) to Class IV (worst).
  Record any change from baseline in percentage of patients in NYHA class IV/III/II class over the course of 12 weeks.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | From baseline to 12 weeks of treatment
  Any changes from baseline KCCQ compared to after 12 weeks of treatment Where "No limits" is the best outcome and "Severely limited" is the worst outcome.
Time to resolution of clinical symptoms | From baseline to 12 weeks of treatment
  chest pain, arrhythmias, shortness of breath
Changes in inflammatory and biomarker hs-troponin (nh/ml) | From baseline to 12 weeks of treatment
  Patients with myocarditis present with abnormal (very high) values in inflammatory and biomarkers.
  The investigators are trying to determine if CardiolRx normalizes them faster than placebo.
Changes in inflammatory and biomarkers NT-proBNP (pg/ml), TNF-alpha (pg/ml), IL-1 beta (pg/ml) and IL-6 (pg/ml) | From baseline to 12 weeks of treatment
  Patients with myocarditis present with abnormal (very high) values in inflammatory and biomarkers.
  The investigators are trying to determine if CardiolRx normalizes them faster than placebo.
Changes in inflammatory and biomarkers hs-CRP (mg/l), and ferritin (mg/l) | From baseline to 12 weeks of treatment
  Patients with myocarditis present with abnormal (very high) values in inflammatory and biomarkers.
  The investigators are trying to determine if CardiolRx normalizes them faster than placebo.
Changes in inflammatory and biomarker IL-10 (ng/ml) | From baseline to 12 weeks of treatment
  Patients with myocarditis present with abnormal (very high) values in inflammatory and biomarkers.
  The investigators are trying to determine if CardiolRx normalizes them faster than placebo.
Normalization of prognostically important ECG changes | From baseline to 12 weeks of treatment
  Time to normalization of normalization of PR interval
Normalization of prognostically important ECG changes | From baseline to 12 weeks of treatment
  Time to normalization of normalization of QRS duration
Normalization of prognostically important ECG changes | From baseline to 12 weeks of treatment
  Time to normalization of normalization of ST/T wave changes

CONTACTS AND LOCATIONS:
Overall Officials: Dennis McNamara, MD, Study Chair — University of Pittsburgh
Locations (37):
- United States (6):
  - MedStar Heart and Vascular Institute, Washington D.C., District of Columbia
  - Massachusetts General Hospital site, Boston, Massachusetts
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia
- Brazil (14):
  - Nupec-Orizonti, Belo Horizonte, Minas Gerais
  - PUC trials, Curitiba, Paraná
  - Complexo Hospitalar de Niterói, Niterói, Rio de Janeiro
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul
  - Hospital Nove de Julho, São Paulo, São Paulo
  - Hospital Felicio Rocho - Fundação Felice Rosso, Belo Horizonte
  - Hospital Angelina Caron, Campina Grande do Sul
  - Hospital São Lucas, Porto Alegre
  - Instituto D´Or de Pesquisa e Ensino, Rio de Janeiro
  - Hospital Pró-Cardíaco, Rio de Janeiro
  - Hospital Regional de São José, São José
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo
  - Instituto do Coração - InCor, São Paulo
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - McGill University Health Centre, Montreal, Quebec
- France (10):
  - Hopital Louis Pradel Hospices Civils de Lyon, Bron
  - CHU de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Hôpital Lariboisière - Département de Cardiologie, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Hôpital européen Georges-Pompidou, Paris
  - Institut de Cardiologie hopital Pitié Salpêtrière, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hôpital Foch, Suresnes
  - Chu Rangueil, Toulouse
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Shaare Zedek Medical Center, Jerusalem
  - Beilinson Hospital, Rabin medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center (Ichilov), Tel Aviv
  - Shamir Medical Center (Assaf Harofeh), Zrifin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee WS, Erdelyi K, Matyas C, Mukhopadhyay P, Varga ZV, Liaudet L, Hasku G, Cihakova D, Mechoulam R, Pacher P. Cannabidiol Limits T Cell-Mediated Chronic Autoimmune Myocarditis: Implications to Autoimmune Disorders and Organ Transplantation. Mol Med. 2016 Sep;22:136-146. doi: 10.2119/molmed.2016.00007. Epub 2016 Jan 8. PMID 26772776